CLINICAL TRIAL: NCT02375243
Title: Use of Dexmedetomidine in Children Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bambino Gesù Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Cristiana Garisto, physician, Bambino Gesù Hospital and Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 942LB
Record Dates: First submitted 2014-10-25; First posted 2015-03-02 (Estimated); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Deep Sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cases (Experimental): children who receive midazolam 0.05 mg/kg/h + morphine 10 mcg/kg/h + dexmedetomidne 0.5 mcg/kg/h. Midazolam in administered until extubation, while morphine and dexmedetomidine are administered until removal of surgical drains.
  Interventions: Drug: dexmedetomidine
- controls (No Intervention): standard care: children who receive midazolam 0.1 mg/kg/h + morphine 20 mcg/kg/h. Midazolam in administered until extubation, while morphine is administered until removal of surgical drains.

INTERVENTIONS:
Drug: dexmedetomidine — dexmedetomidine continous infusion 0.5 mcg/kg/h
  Other Names: dexdor
  Arms: cases

SUMMARY:
The aim of the study is to evaluate the efficacy of dexmedetomidine in reducing the need for sedatives and analgesics in the immediate post-operative period in children who underwent surgical correction of complex congenital heart disease

DETAILED DESCRIPTION:
The hypothesis the investigators want to verify is that the reduced administration of sedative drugs (opioids and benzodiazepines) in children undergoing cardiac surgery, reduces the side effects of the drugs themselves, such as respiratory depression (reduction of mechanical ventilation) and the onset of withdrawal symptoms while maintaining an adequate analgo-sedation.

The study is an unblinded randomized controlled study. It will involve 60 children aged > 1 and < 24 months sedated and mechanically ventilated after corrective or palliative surgery of congenital heart disease on cardiopulmonary bypass with Aristotle score > 8.

Dexmedetomidine infusion will be started upon arrival in the CICU and continued until the time of discontinuation of morphine.

ELIGIBILITY:
Inclusion Criteria: age < 24 months but > 30 days, Aristotle score >8, elective procedures in cardiopulmonary bypass -

Exclusion Criteria: atrioventricular block prior to the start of infusion; vasoactive inotropic score on arrival to the CICU>30; brain malformations orbone, muscle or neuromuscolar disease; pleural effusion or pneumothorax prior to the study; hepatic or renal failure

-

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
mechanical ventilation time | participants will be followed for the duration of ICU stay, an expected average of 5 days
  To evaluate the efficacy of dexmedetomidine, administered in combination with midazolam and morphine, in reducing the time of mechanical ventilation, due to lower consumption of opioids and hypnotics and subsequent reduction of respiratory depression

SECONDARY OUTCOMES:
analgo-sedation level | participants will be followed for the duration of ICU stay, an expected average of 5 days
  efficient analgo-sedation guaranteed by the effectiveness of opioids and benzodiazepines with dexmedetomidine by using the Comfort scale and measuring the total amount of opioids and benzodiazepines received in the two groups.
withdrawal symptoms | participants will be followed for the duration of ICU stay, an expected average of 5 days
  onset of withdrawal symptoms due to abstinence from opioids and benzodiazepines evaluated using Sophia Observation withdrawal Symptoms scale in patients who received a continuous infusion for at least 72 hours
safety of dexmedetomidine infusion as a measure of systemic pressure decrease | participants will be followed for the duration of ICU stay, an expected average of 5 days
  assessment of the safety of dexmedetomidine infusion in light of hemodynamic changes induced by the drug (hypotension will be considered a reduction of > 20% of the mean arterial pressure, bradycardia a reduction in heart rate >20% of baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paola Cogo, doctor, Study Chair — Bambino Gesù Children Hospital
Locations (1):
- Bambino Gesù Children's Hospital, Rome, Rome, Italy